CLINICAL TRIAL: NCT01202279
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of the Safety and Efficacy of Mucinex D for Symptomatic Therapy in Patients With Acute Upper Respiratory Tract Who Seek Treatment
Brief Title: Safety and Efficacy Study of Guaifenesin and Pseudoephedrine for Symptomatic Therapy to Treat Acute RTI
Acronym: Wait and See
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reckitt Benckiser Inc. (Industry)
Responsible Party: Sponsor
Organization: Reckitt Benckiser LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-MUCD-001
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Acute Upper Respiratory Track Infection
Keywords: Acute Upper Respiratory Track Infection Who Seek Treatment
MeSH Terms: interventions — Guaifenesin; Amiloride; Acetylcysteine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mucinex D (Active Comparator): Mucinex D (1200 mg guaifenesin and 120 mg pseudoephedrine HCl) extended release bilayer tablet twice a day (bid) with a full glass of water for 7 days
  Interventions: Drug: Guaifenesin
- Placebo (Placebo Comparator): Placebo given bid with a full glass of water for 7 days
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: Guaifenesin — 1200 mg guaifenesin and 120 mg pseudoephedrine HCl bid for 7 days
  Other Names: Mucinex D; Mucinex; Pseudoephedrine
  Arms: Mucinex D
Device: Placebo — Placebo bid for 7 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment with Mucinex D lowers the use of antibiotics in the treatment of upper respiratory infection when compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 75 yrs of age presenting at a clinical site with symptoms diagnostic for an acute upper respiratory tract infection within the last 5 days

Exclusion Criteria:

* patients who had chronic, recurring respiratory signs and symptoms due to conditions such as chronic allergic rhinitis, chronic sinusitis or chronic bronchitis which in the investigator's opinion, confounded interpretation of symptom ratings for the acute upper respiratory infection. Also excluded were patients with a fever greater than 101 degrees F.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Clinical Research Advantage, Inc., Mesa, Arizona
  - Med Center, Carmichael, California
  - Research Center of Fresno, 3636 N. First Street, Suite 141, Fresno, California
  - Coastal Medical Research Group, Inc., 47 Santa Rosa Street, San Luis Obispo, California
  - Coastal Connecticut Research, LLC, 342 Montauk Avenue, New London, Connecticut
  - Glasgow Family Practice, Newark, Delaware
  - Koch Family Medicine, 81A E. Queenwood Road, Morton, Illinois
  - Sterling Research Group, Ltd., 650 Sprucewood Lane, Erlanger, Kentucky
  - Clinical Associates Research, 750 Main Street, Suite 310, Reisterstown, Maryland
  - Park Place Family Practice & Internal Medicine, Taylor, Michigan
  - Immedicenter, Bloomfield, New Jersey
  - Peters Medical Research, High Point, North Carolina
  - (Piedmont Medical Research Assoc., Inc. d/b/a), Crescent Medical Research, Salisbury, North Carolina
  - Parsons Avenue Medical Clinic, Columbus, Ohio
  - Legacy Clinical Research, LLC, 1204 W. Willow Road, Suite B, Enid, Oklahoma
  - Integrated Medical Research, PC, Ashland, Oregon
  - Harleysville Medical Associates, 176 Main Street, Harleysville, Pennsylvania
  - Kastelic MD & Associates, 322 Warren Street, Suite 300, Johnstown, Pennsylvania
  - Durham Physicians, P.C., Penndel, Pennsylvania
  - Palmetto Medical Research, 180 Wingo Way, Suite 203, Mt. Pleasant, South Carolina
  - TriCities Medical Research, Bristol, Tennessee
  - Village Health Partners, Plano, Texas
  - Independence Family Medicine, 813 Independence Blvd., Suite A, Virginia Beach, Virginia
  - Amherst Family Practice, 1867 Amherst Street, Winchester, Virginia

REFERENCES:
- [Derived] Septimus EJ, Albrecht HH, Solomon G, Shea T, Guenin EP. Extended-Release Guaifenesin/Pseudoephedrine Hydrochloride for Symptom Relief in Support of a Wait-and-See Approach for the Treatment of Acute Upper Respiratory Tract Infections: A Randomized, Double-Blind, Placebo-Controlled Study. Curr Ther Res Clin Exp. 2017 Apr 28;84:54-61. doi: 10.1016/j.curtheres.2017.04.004. eCollection 2017. PMID 28761581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place October 2009 through April 2010. Advertising was not allowed for this study. Patients were seen by a Health Care Provider(HCP) and must have been seeking treatment for symptoms diagnostic for an acute upper respiratory tract infection.
Groups:
- Mucinex D: Mucinex D (1200 mg GGE and 120 mg pseudoephedrine HCl extended release bilayer tablet bid with a full glass of water for 7 days
Period: Overall Study
Arm/Group | Mucinex D | Placebo
Started | 591 | 588
Completed | 554 | 561
Not Completed | 37 | 27
Not completed — Adverse Event | 8 | 6
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 10 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — study compliance | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mucinex D | Placebo | Total
Number analyzed (Participants) | 591 | 588 | 1179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 575 | 575 | 1150
  >=65 years | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (13.7) | 38.8 (13.7) | 38.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 395 | 404 | 799
  Male | 196 | 184 | 380
Region of Enrollment [Number; unit: participants]
  United States | 591 | 588 | 1179

OUTCOME MEASURES:

1. Primary Outcome: Antibiotic Sparing
Description: Number of patients who received an antibiotic
Time Frame: Day 7
Population: Per Protocol Population using Fishers Exact Test.
Measure: Number; unit: Participants
Arm/Group | Mucinex D | Placebo
Number analyzed (Participants) | 510 | 523
Participants | 89 | 121
Statistical Analysis 1: Comparison: Mucinex D vs Placebo; Test type: Superiority or Other; p = 0.025, Fisher Exact

2. Primary Outcome: Change From Baseline in Total Symptom Score of the Wisconsin Upper Respiratory Symptom Survey - 21 (WURSS-21).
Description: WURSS-21 is made up of 21 questions with a scoring from 0 = no symptom to 7 = severe symptom. With a minimum score of 0 to a maximum score of 147.
Time Frame: Baseline and 7 Days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mucinex D | Placebo
Number analyzed (Participants) | 591 | 588
units on a scale | -14.2 (7.71) | -13.4 (7.99)
Statistical Analysis 1: Comparison: Mucinex D vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA

ADVERSE EVENTS:
Time Frame: Upon signing of the informed consent, the patient was requested to report all AEs experienced throughout the duration of their participation in this study. AEs were followed until resolution, stability or until 30 days after last dose of study medication.
Arm/Group | Mucinex D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/593 | 0/591
Other Adverse Events (participants affected / at risk) | 37/593 | 21/591
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex D (N=593) | Placebo (N=591)
Nervousness (Psychiatric disorders) | 7 (7) | 4 (4)
Insomnia (Psychiatric disorders) | 17 (18) | 1 (1)
Headache (Nervous system disorders) | 7 (13) | 14 (21)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less